CLINICAL TRIAL: NCT00277823
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Two Fixed Doses (50 mg, 100 mg) of Desvenlafaxine Sustained-Release Tablets in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Sustained-Release (DVS-SR) in Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-332
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Adult; Outpatients
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Drug: DVS-SR 50 mg
Drug: DVS-SR 100 mg
Drug: Placebo

SUMMARY:
The purpose of this study is to compare the antidepressant efficacy, safety, and tolerability of DVS-SR in subjects receiving daily doses of 50 mg or 100 mg of DVS-SR versus subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive disorder
* Must be able to swallow tablets
* Must be at least 18 years of age.

Exclusion Criteria:

* Clinical diagnosis of other psychiatric disorders
* Significant risk of suicide
* Unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2006-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare the antidepressant efficacy, safety, and tolerability of DVS-SR in subjects receiving daily doses of 50 mg or 100 mg of DVS SR versus subjects receiving placebo.

SECONDARY OUTCOMES:
Additional objectives include testing both general and functional quality-of-life outcomes and satisfaction with therapy reported by the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (24):
- United States (24):
  - Beverly Hills, California
  - Northridge, California
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Miami, Florida
  - St. Petersburg, Florida
  - Marietta, Georgia
  - Smyrna, Georgia
  - Libertyville, Illinois
  - New Orleans, Louisiana
  - Farmington Hills, Michigan
  - Clementon, New Jersey
  - Moorestown, New Jersey
  - New York, New York
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Salt Lake City, Utah
  - Seattle, Washington
  - Brown Deer, Wisconsin

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Soares CN, Endicott J, Boucher M, Fayyad RS, Guico-Pabia CJ. Predictors of functional response and remission with desvenlafaxine 50 mg/d in patients with major depressive disorder. CNS Spectr. 2014 Dec;19(6):519-27. doi: 10.1017/S1092852914000066. Epub 2014 Feb 26. PMID 24571916
- [Derived] Liebowitz MR, Manley AL, Padmanabhan SK, Ganguly R, Tummala R, Tourian KA. Efficacy, safety, and tolerability of desvenlafaxine 50 mg/day and 100 mg/day in outpatients with major depressive disorder. Curr Med Res Opin. 2008 Jul;24(7):1877-90. doi: 10.1185/03007990802161923. Epub 2008 May 27. PMID 18507895